CLINICAL TRIAL: NCT02545868
Title: A Phase IIIB, Multicenter, Randomized, Parallel-Group, Open-Label Study to Evaluate the Effects of Ocrelizumab on Immune Responses in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: A Study to Evaluate the Effects of Ocrelizumab on Immune Responses In Participants With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BN29739; 2015-001357-32 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Influenza Vaccines; ocrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: OCR + Vaccines (Experimental): Participants will receive dual infusion of OCR 300 milligrams (mg) on Day 1 and then on Day 15, and then participants will further receive immunization course (TT-containing adsorbed vaccine, 23-PPV either unboosted or boosted with 13-PCV, influenza vaccine, and repeated administration with KLH) at 12 weeks post-OCR treatment until Week 24. Participants who complete the 24-week immunization study period will have the option for retreatment with a single infusion of 600 mg OCR on Day 169 and subsequent single infusions (600 mg OCR) at intervals of 24 weeks. Participants who have received one or more infusions of OCR will enter the 48-week safety follow-up period.
  Interventions: Biological: 23-PPV; Biological: 13-PCV Booster; Biological: Influenza Vaccine; Biological: KLH; Drug: OCR; Biological: TT Vaccine
- Group B: Vaccines (Optional OCR in Extension) (Other): Participants will receive immunizations (TT-containing adsorbed vaccine, 23-PPV, influenza vaccine, and repeated administration with KLH) on Day 1 until Week 12 of the immunization period.
  Interventions: Biological: 23-PPV; Biological: Influenza Vaccine; Biological: KLH; Drug: OCR; Biological: TT Vaccine

INTERVENTIONS:
Biological: 23-PPV — The 23-PPV vaccine will be given as a 0.5-milliliter (mL) intramuscular (IM) injection in the deltoid muscle on Day 112 (Group A) or Day 28 (Group B).
Biological: 13-PCV Booster — The 13-PCV booster will be given as an IM injection in the deltoid muscle on Day 140 (select participants in Group A).
  Arms: Group A: OCR + Vaccines
Biological: Influenza Vaccine — The influenza vaccine will be given as an IM injection in the deltoid muscle at any time between Day 85 and Day 144 (select participants in Group A) or any time between Day 1 and Day 85 (Group B).
Biological: KLH — KLH will be given as a 1-mg subcutaneous (SC) injection on Days 84, 112, and 140 (Group A) or Days 1, 28, and 56 (Group B).
Drug: OCR — OCR will be given as an intravenous (IV) infusion at a dose of 600 mg, with the first dose given as two infusions of 300mg 14 days apart, according to the specifications described in the corresponding Group A and Group B arms.
  Other Names: RO4964913, PRO70769, rhuMAb 2H7
Biological: TT Vaccine — The TT-containing adsorbed vaccine will be given as a 0.5-mL IM injection in the deltoid muscle on Day 85 (Group A) or Day 1 (Group B).

SUMMARY:
This multicenter, randomized, open-label study will evaluate the immune response to vaccines (tetanus toxoid [TT]-containing adsorbed vaccine, 23-valent pneumococcal polysaccharide vaccine [23-PPV] either unboosted or boosted with 13-valent pneumococcal conjugate vaccine [13-PCV], influenza vaccine, keyhole limpet hemocyanin [KLH]) after administration of a dose of ocrelizumab (OCR) in participants with relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RMS in accordance with the revised McDonald criteria
* Received at least one previous immunization against TT or tetanus and diphtheria (DT/Td) or tetanus, diphtheria, and acellular pertussis (DTaP/Tdap)
* Expanded Disability Status Scale (EDSS) at Screening from 0 to 5.5 points, inclusive
* For sexually active female participants of reproductive potential, use of reliable means of contraception

Exclusion Criteria:

* Contraindications for or intolerance to oral or IV corticosteroids, including IV methylprednisolone, according to the country label
* Known presence of other neurologic disorders
* Treatment with any investigational agent within 24 weeks of screening or 5 half-lives of the investigational drug, whichever is longer, or treatment with any experimental procedure for multiple sclerosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (20):
  - North Central Neurology Associates, Cullman, Alabama
  - Territory Neurology and Research Institute, Tucson, Arizona
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Scripps Clinic, La Jolla, California
  - University of Miami School of Medicine; Dept. of Neurology Movement Disorder Center, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Mercy Hospital St. Louis / Mercy Clinic Neurology, Chesterfield, Missouri
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - Staten Island Univ Hospital, Staten Island, New York
  - Neurology Associates PA, Hickory, North Carolina
  - Ohio Health Research Institute Grant Medical Center, Columbus, Ohio
  - MDH Research LLC, Westerville, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - Neurology Clinic PC, Cordova, Tennessee
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Rocky Mountain MS Clinic, Salt Lake City, Utah
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia Hospital; Division of Neurology, Vancouver, British Columbia

REFERENCES:
- [Derived] Bar-Or A, Calkwood JC, Chognot C, Evershed J, Fox EJ, Herman A, Manfrini M, McNamara J, Robertson DS, Stokmaier D, Wendt JK, Winthrop KL, Traboulsee A. Effect of ocrelizumab on vaccine responses in patients with multiple sclerosis: The VELOCE study. Neurology. 2020 Oct 6;95(14):e1999-e2008. doi: 10.1212/WNL.0000000000010380. Epub 2020 Jul 29. PMID 32727835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited participants with relapsing forms of multiple sclerosis in 2 countries from 27 October 2015 to 14 February 2017.
Pre-assignment Details: A total of 122 participants were screened of which 102 participants were randomized.
Groups:
- Group A1: Participants received dual infusion of OCR 300 mg on Day 1 and then on Day 15, and then participants further received immunization course: TT containing adsorbed vaccine, 23-PPV boosted with 13-PCV and repeated administration with KLH at 12 weeks post-OCR treatment until Week 24.
- Group A2: Participants received dual infusion of OCR 300 mg on Day 1 and then on Day 15, and then participants further received immunization course: TT containing adsorbed vaccine, 23-PPV, influenza vaccine, and repeated administration with KLH at 12 weeks post-OCR treatment until Week 24.
- Group B: Participants received immunizations (TT-containing adsorbed vaccine, 23-PPV, influenza vaccine, and repeated administration with KLH) on Day 1 until Week 12 of the immunization period.
Period: Overall Study
Arm/Group | Group A1 | Group A2 | Group B
Started | 33 | 35 | 34
Completed | 2 | 1 | 0
Not Completed | 31 | 34 | 34
Not completed — Lack of Efficacy | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 5 | 1
Not completed — Non-compliance | 1 | 1 | 1
Not completed — Treatment change | 21 | 19 | 22
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Withdrawal by Subject | 6 | 7 | 9

BASELINE CHARACTERISTICS:
Population: Observed Cases (OC) Population was defined as all randomized participants who completed the ISP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A1 | Group A2 | Group B | Total
Number analyzed (Participants) | 33 | 35 | 34 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (8.0) | 39.3 (9.7) | 41.4 (7.9) | 40.3 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 27 | 72
  Male | 12 | 11 | 7 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 2 | 2 | 2 | 6
  Ethnicity: Not Hispanic or Latino | 29 | 30 | 32 | 91
  Ethnicity: Not reported | 1 | 1 | 0 | 2
  Ethnicity: Unknown | 1 | 2 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 0 | 2 | 3
  Race: Black or African American | 0 | 3 | 2 | 5
  Race: White | 32 | 32 | 30 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Positive Response to TT Vaccine Measured 8 Weeks After TT Vaccine
Description: For participants with pre-vaccination tetanus antibody titers < 0.1 IU/mL, a positive response was defined as an antibody titer >/= 0.2 IU/mL measured 8 weeks after vaccination. For participants with pre-vaccination tetanus antibody titers >/= 0.1 IU/mL, a positive response was defined as at least a 4-fold increase in antibody titers measured 8 weeks after vaccination compared with pre-vaccination levels.
Time Frame: 8 weeks after TT vaccine
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Groups:
- Group A (A1 + A2): Participants received dual infusion of ocrelizumab (OCR) 300 milligrams (mg) on Days 1 and 15, and then further received the following immunization course during the period from Week 12 to Week 24: tetanus toxoid (TT) containing adsorbed vaccine, 23-valent pneumococcal polysaccharide vaccine (23-PPV) and repeated administration with keyhole limpet hemocyanin (KLH). In addition, only Group A1 received 13-valent pneumococcal conjugate vaccine (13-PCV, booster to 23-PPV) and only Group A2 received influenza vaccine.
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants | 23.9 | 54.5
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Difference in positive response, Group A minus Group B; Test type: Superiority; normal distribution approximation = -30.7, 95% CI 2-sided [-50.5 to -10.8]

2. Secondary Outcome: Percentage of Participants With Positive Response to TT Vaccine Measured 4 Weeks After TT Vaccine
Description: For participants with pre-vaccination tetanus antibody titers < 0.1 IU/mL, a positive response was defined as an antibody titer >/= 0.2 IU/mL measured 4 weeks after vaccination. For participants with pre-vaccination tetanus antibody titers >/= 0.1 IU/mL, a positive response was defined as at least a 4-fold increase in antibody titers measured 4 weeks after vaccination compared with pre-vaccination levels.
Time Frame: 4 weeks after TT vaccine
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Groups:
- Group A (A1 + A2): Participants received dual infusion of OCR 300 mg on Days 1 and 15, and then further received the following immunization course during the period from Week 12 to Week 24: TT containing adsorbed vaccine, 23-PPV and repeated administration with KLH. In addition, only Group A1 received 13-valent pneumococcal conjugate vaccine (13-PCV, booster to 23-PPV) and only Group A2 received influenza vaccine.
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants | 24.2 | 60.6
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Difference in positive response, Group A minus Group B; Test type: Superiority; normal distribution approximation = -36.4, 95% CI 2-sided [-56.0 to -16.7]

3. Secondary Outcome: Percentage of Participants With Tetanus Antibody Titer >/=0.2 IU/mL or 2-Fold Increase in Tetanus Antibody Titers
Description: For participants with pre-vaccination tetanus antibody titers < 0.1 IU/mL, a positive response was defined as an antibody titer >/= 0.2 IU/mL measured 4 weeks after vaccination. For participants with pre-vaccination tetanus antibody titers >/= 0.1 IU/mL, a positive response was defined as at least a 2-fold increase in antibody titers measured 4 weeks after vaccination compared with pre-vaccination levels.
Time Frame: 4 weeks after TT vaccine
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants | 40.9 | 87.9
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Difference in positive response, Group A minus Group B; Test type: Superiority; normal distribution approximation = -47.0, 95% CI 2-sided [-63.2 to -30.7]

4. Secondary Outcome: Mean Levels of Anti-Tetanus Antibody
Description: Anti-tetanus antibody levels were assessed by enzyme-linked immunosorbent assay (ELISA).
Time Frame: Immediately prior to and at 4 and 8 weeks after TT vaccine
Population: OC population included all randomized participants who completed the ISP.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
IU/mL
  Pre-Vaccination: number analyzed (Participants) | 67 | 34
  Pre-Vaccination | 1.680 [1.275 to 2.214] | 2.147 [1.612 to 2.859]
  4 weeks after TT vaccine: number analyzed (Participants) | 67 | 33
  4 weeks after TT vaccine | 4.132 [3.373 to 5.061] | 12.157 [9.498 to 15.560]
  8 weeks after TT vaccine: number analyzed (Participants) | 68 | 33
  8 weeks after TT vaccine | 3.743 [3.048 to 4.596] | 9.812 [7.842 to 12.277]

5. Secondary Outcome: Mean Levels of Anti-KLH Antibody: Immunoglobulin (Ig) G
Description: Anti-KLH antibody levels were assessed by ELISA.
Time Frame: Immediately prior to first KLH administration and 4, 8, and 12 weeks after first KLH administration
Population: OC population included all randomized participants who completed the ISP.
Measure: Geometric Mean (95% Confidence Interval); unit: titer units
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
titer units
  Immediately prior to first KLH administration | 274 [213 to 354] | 235 [180 to 308]
  4 weeks after first KLH administration | 384 [285 to 517] | 1086 [769 to 1534]
  8 weeks after first KLH administration | 2916 [1998 to 4253] | 17737 [12441 to 25287]
  12 weeks after first KLH administration: number analyzed (Participants) | 66 | 34
  12 weeks after first KLH administration | 5298 [3794 to 7397] | 60270 [43557 to 83396]

6. Secondary Outcome: Mean Levels of Anti-KLH Antibody: Ig M
Description: Anti-KLH antibody levels were assessed by ELISA.
Time Frame: Immediately prior to first KLH administration and 4, 8, and 12 weeks after first KLH administration
Population: OC population included all randomized participants who completed the ISP.
Measure: Geometric Mean (95% Confidence Interval); unit: titer units
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
titer units
  Immediately prior to first KLH administration: number analyzed (Participants) | 67 | 34
  Immediately prior to first KLH administration | 100 [82 to 122] | 130 [101 to 168]
  4 weeks after first KLH administration: number analyzed (Participants) | 67 | 34
  4 weeks after first KLH administration | 124 [100 to 155] | 217 [158 to 298]
  8 weeks after first KLH administration | 361 [273 to 478] | 1086 [797 to 1481]
  12 weeks after first KLH administration: number analyzed (Participants) | 66 | 34
  12 weeks after first KLH administration | 372 [286 to 483] | 1883 [1405 to 2524]

7. Secondary Outcome: Percentage of Participants With Positive Response Against Individual Pneumococcal Serotypes in 23-PPV
Description: Positive response against a serotype was defined as a 2-fold increase in anti-pneumococcal antibody level or greater than (>) 1 microgram per milliliter (mcg/mL) rise compared with pre-vaccination levels.
Time Frame: 4 weeks after 23-PPV
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants
  Serotype 1: number analyzed (Participants) | 67 | 34
  Serotype 1 | 49.3 | 100.0
  Serotype 2: number analyzed (Participants) | 67 | 34
  Serotype 2 | 53.7 | 97.1
  Serotype 3: number analyzed (Participants) | 67 | 34
  Serotype 3 | 34.3 | 82.4
  Serotype 4: number analyzed (Participants) | 67 | 34
  Serotype 4 | 28.4 | 91.2
  Serotype 5: number analyzed (Participants) | 67 | 34
  Serotype 5 | 40.3 | 94.1
  Serotype 6B: number analyzed (Participants) | 67 | 34
  Serotype 6B | 47.8 | 85.3
  Serotype 7F: number analyzed (Participants) | 67 | 34
  Serotype 7F | 32.8 | 91.2
  Serotype 8: number analyzed (Participants) | 67 | 34
  Serotype 8 | 64.2 | 97.1
  Serotype 9N: number analyzed (Participants) | 67 | 34
  Serotype 9N | 41.8 | 88.2
  Serotype 9V: number analyzed (Participants) | 67 | 34
  Serotype 9V | 50.7 | 91.2
  Serotype 10A: number analyzed (Participants) | 67 | 34
  Serotype 10A | 28.4 | 91.2
  Serotype 11A: number analyzed (Participants) | 67 | 34
  Serotype 11A | 29.9 | 82.4
  Serotype 12F: number analyzed (Participants) | 67 | 34
  Serotype 12F | 20.9 | 76.5
  Serotype 14: number analyzed (Participants) | 67 | 34
  Serotype 14 | 62.7 | 88.2
  Serotype 15B: number analyzed (Participants) | 67 | 34
  Serotype 15B | 40.3 | 88.2
  Serotype 17F: number analyzed (Participants) | 67 | 34
  Serotype 17F | 31.3 | 88.2
  Serotype 18C: number analyzed (Participants) | 67 | 34
  Serotype 18C | 38.8 | 91.2
  Serotype 19A: number analyzed (Participants) | 67 | 34
  Serotype 19A | 41.8 | 88.2
  Serotype 19F: number analyzed (Participants) | 67 | 34
  Serotype 19F | 32.8 | 85.3
  Serotype 20: number analyzed (Participants) | 67 | 34
  Serotype 20 | 20.9 | 82.4
  Serotype 22F: number analyzed (Participants) | 67 | 34
  Serotype 22F | 34.3 | 91.2
  Serotype 23F: number analyzed (Participants) | 67 | 34
  Serotype 23F | 43.3 | 76.5
  Serotype 33F: number analyzed (Participants) | 67 | 34
  Serotype 33F | 46.3 | 94.1
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Serotype 1; Test type: Superiority; Normal Distribution Approximation = -50.7, 95% CI 2-sided [-62.7 to -38.8]
Statistical Analysis 2: Comparison: Group A (A1 + A2) vs Group B; Serotype 2; Test type: Superiority; Normal Distribution Approximation = -43.3, 95% CI 2-sided [-56.5 to -30.1]
Statistical Analysis 3: Comparison: Group A (A1 + A2) vs Group B; Serotype 3; Test type: Superiority; Normal Distribution Approximation = -48.0, 95% CI 2-sided [-65.2 to -30.9]
Statistical Analysis 4: Comparison: Group A (A1 + A2) vs Group B; Serotype 4; Test type: Superiority; Normal Distribution Approximation = -62.8, 95% CI 2-sided [-77.2 to -48.4]
Statistical Analysis 5: Comparison: Group A (A1 + A2) vs Group B; Serotype 5; Test type: Superiority; Normal Distribution Approximation = -53.8, 95% CI 2-sided [-68.0 to -39.7]
Statistical Analysis 6: Comparison: Group A (A1 + A2) vs Group B; Serotype 6B; Test type: Superiority; Normal Distribution Approximation = -37.5, 95% CI 2-sided [-54.4 to -20.7]
Statistical Analysis 7: Comparison: Group A (A1 + A2) vs Group B; Serotype 7F; Test type: Superiority; Normal Distribution Approximation = -58.3, 95% CI 2-sided [-73.1 to -43.6]
Statistical Analysis 8: Comparison: Group A (A1 + A2) vs Group B; Serotype 8; Test type: Superiority; Normal Distribution Approximation = -32.9, 95% CI 2-sided [-45.7 to -20.1]
Statistical Analysis 9: Comparison: Group A (A1 + A2) vs Group B; Serotype 9N; Test type: Superiority; Normal Distribution Approximation = -46.4, 95% CI 2-sided [-62.5 to -30.4]
Statistical Analysis 10: Comparison: Group A (A1 + A2) vs Group B; Serotype 9V; Test type: Superiority; Normal Distribution Approximation = -40.4, 95% CI 2-sided [-55.7 to -25.1]
Statistical Analysis 11: Comparison: Group A (A1 + A2) vs Group B; Serotype 10A; Test type: Superiority; Normal Distribution Approximation = -62.8, 95% CI 2-sided [-77.2 to -48.4]
Statistical Analysis 12: Comparison: Group A (A1 + A2) vs Group B; Serotype 11A; Test type: Superiority; Normal Distribution Approximation = -52.5, 95% CI 2-sided [-69.4 to -35.6]
Statistical Analysis 13: Comparison: Group A (A1 + A2) vs Group B; Serotype 12F; Test type: Superiority; Normal Distribution Approximation = -55.6, 95% CI 2-sided [-72.8 to -38.3]
Statistical Analysis 14: Comparison: Group A (A1 + A2) vs Group B; Serotype 14; Test type: Superiority; Normal Distribution Approximation = -25.5, 95% CI 2-sided [-41.4 to -9.7]
Statistical Analysis 15: Comparison: Group A (A1 + A2) vs Group B; Serotype 15B; Test type: Superiority; Normal Distribution Approximation = -47.9, 95% CI 2-sided [-63.9 to -32.0]
Statistical Analysis 16: Comparison: Group A (A1 + A2) vs Group B; Serotype 17F; Test type: Superiority; Normal Distribution Approximation = -56.9, 95% CI 2-sided [-72.4 to -41.4]
Statistical Analysis 17: Comparison: Group A (A1 + A2) vs Group B; Serotype 18C; Test type: Superiority; Normal Distribution Approximation = -52.4, 95% CI 2-sided [-67.4 to -37.3]
Statistical Analysis 18: Comparison: Group A (A1 + A2) vs Group B; Serotype 19A; Test type: Superiority; Normal Distribution Approximation = -46.4, 95% CI 2-sided [-62.5 to -30.4]
Statistical Analysis 19: Comparison: Group A (A1 + A2) vs Group B; Serotype 19F; Test type: Superiority; Normal Distribution Approximation = -52.5, 95% CI 2-sided [-68.8 to -36.1]
Statistical Analysis 20: Comparison: Group A (A1 + A2) vs Group B; Serotype 20; Test type: Superiority; Normal Distribution Approximation = -61.5, 95% CI 2-sided [-77.5 to -45.4]
Statistical Analysis 21: Comparison: Group A (A1 + A2) vs Group B; Serotype 22F; Test type: Superiority; Normal Distribution Approximation = -56.8, 95% CI 2-sided [-71.7 to -42.0]
Statistical Analysis 22: Comparison: Group A (A1 + A2) vs Group B; Serotype 23F; Test type: Superiority; Normal Distribution Approximation = -33.2, 95% CI 2-sided [-51.7 to -14.6]
Statistical Analysis 23: Comparison: Group A (A1 + A2) vs Group B; Serotype 33F; Test type: Superiority; Normal Distribution Approximation = -47.8, 95% CI 2-sided [-62.2 to -33.5]

8. Secondary Outcome: Percentage of Participants With Positive Response Against >/=2 Pneumococcal Serotypes
Description: Positive response against a serotype was defined as a 2-fold increase in anti-pneumococcal antibody level or > 1 mcg/mL rise compared with pre-vaccination levels.
Time Frame: 4 weeks after 23-PPV
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants | 86.6 | 100.0
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Test type: Superiority; Normal Distribution Approximation = -13.4, 95% CI 2-sided [-21.6 to -5.3]

9. Secondary Outcome: Percentage of Participants With Positive Response Against >/=12 Pneumococcal Serotypes
Description: as for outcome 8
Time Frame: 4 weeks after 23-PPV
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants | 37.3 | 97.1
Statistical Analysis 1: Comparison: Group A (A1 + A2) vs Group B; Test type: Superiority; Normal Distribution Approximation = -59.7, 95% CI 2-sided [-72.6 to -46.8]

10. Secondary Outcome: Mean Levels of Anti-Pneumococcal Antibody
Description: Serotype-specific antibody levels (IgG) were assessed by bead-based multi-analyte immunodetection (MAID).
Time Frame: Immediately prior to and 4 weeks after 23-PPV
Population: OC population included all randomized participants who completed the ISP.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
mcg/mL
  Immediately prior to 23-PPV: Serotype : 1: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 1 | 0.94 [0.71 to 1.26] | 1.02 [0.71 to 1.46]
  Immediately prior to 23-PPV: Serotype : 2: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 2 | 1.12 [0.85 to 1.47] | 1.25 [0.93 to 1.69]
  Immediately prior to 23-PPV: Serotype : 3: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 3 | 1.10 [0.81 to 1.50] | 0.95 [0.66 to 1.36]
  Immediately prior to 23-PPV: Serotype : 4: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 4 | 0.68 [0.41 to 1.13] | 0.59 [0.40 to 0.88]
  Immediately prior to 23-PPV: Serotype : 5: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 5 | 0.96 [0.72 to 1.27] | 1.31 [0.91 to 1.89]
  Immediately prior to 23-PPV: Serotype : 6B: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 6B | 0.84 [0.63 to 1.11] | 0.92 [0.60 to 1.39]
  Immediately prior to 23-PPV: Serotype : 7F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 7F | 0.89 [0.72 to 1.10] | 0.94 [0.70 to 1.27]
  Immediately prior to 23-PPV: Serotype : 8: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 8 | 0.92 [0.68 to 1.23] | 0.91 [0.59 to 1.38]
  Immediately prior to 23-PPV: Serotype : 9N: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 9N | 0.74 [0.55 to 1.01] | 1.06 [0.68 to 1.64]
  Immediately prior to 23-PPV: Serotype : 9V: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 9V | 0.79 [0.55 to 1.13] | 0.74 [0.50 to 1.11]
  Immediately prior to 23-PPV: Serotype : 10A: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 10A | 0.88 [0.66 to 1.17] | 0.96 [0.73 to 1.26]
  Immediately prior to 23-PPV: Serotype : 11F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 11F | 1.09 [0.81 to 1.45] | 1.03 [0.69 to 1.52]
  Immediately prior to 23-PPV: Serotype : 12F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 12F | 0.79 [0.46 to 1.36] | 0.54 [0.35 to 0.83]
  Immediately prior to 23-PPV: Serotype : 14: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 14 | 1.33 [0.97 to 1.84] | 1.09 [0.71 to 1.68]
  Immediately prior to 23-PPV: Serotype : 15B: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 15B | 0.82 [0.68 to 1.00] | 1.18 [0.73 to 1.92]
  Immediately prior to 23-PPV: Serotype : 17F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 17F | 0.89 [0.70 to 1.14] | 1.05 [0.75 to 1.48]
  Immediately prior to 23-PPV: Serotype : 18C: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 18C | 1.08 [0.83 to 1.41] | 1.14 [0.79 to 1.64]
  Immediately prior to 23-PPV: Serotype : 19A: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 19A | 1.58 [1.14 to 2.20] | 2.09 [1.26 to 3.46]
  Immediately prior to 23-PPV: Serotype : 19F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 19F | 1.09 [0.89 to 1.35] | 1.16 [0.80 to 1.67]
  Immediately prior to 23-PPV: Serotype : 20: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 20 | 1.71 [1.27 to 2.29] | 1.29 [0.89 to 1.87]
  Immediately prior to 23-PPV: Serotype : 22F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 22F | 0.73 [0.55 to 0.97] | 0.82 [0.55 to 1.20]
  Immediately prior to 23-PPV: Serotype : 23F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 23F | 0.72 [0.56 to 0.93] | 0.96 [0.66 to 1.41]
  Immediately prior to 23-PPV: Serotype : 33F: number analyzed (Participants) | 67 | 34
  Immediately prior to 23-PPV: Serotype : 33F | 0.96 [0.76 to 1.22] | 0.67 [0.52 to 0.85]
  4 weeks after 23-PPV: Serotype : 1 | 1.31 [1.03 to 1.67] | 11.58 [7.72 to 17.38]
  4 weeks after 23-PPV: Serotype : 2 | 1.79 [1.38 to 2.30] | 9.41 [6.80 to 13.01]
  4 weeks after 23-PPV: Serotype : 3 | 1.57 [1.20 to 2.06] | 2.76 [1.72 to 4.42]
  4 weeks after 23-PPV: Serotype : 4 | 1.54 [1.01 to 2.35] | 2.02 [1.32 to 3.08]
  4 weeks after 23-PPV: Serotype : 5 | 1.25 [0.97 to 1.62] | 10.16 [5.69 to 18.15]
  4 weeks after 23-PPV: Serotype : 6B | 1.47 [1.03 to 2.10] | 3.94 [2.12 to 7.33]
  4 weeks after 23-PPV: Serotype : 7F | 1.36 [1.06 to 1.74] | 4.92 [2.99 to 8.09]
  4 weeks after 23-PPV: Serotype : 8 | 1.78 [1.35 to 2.35] | 9.04 [6.42 to 12.73]
  4 weeks after 23-PPV: Serotype : 9N | 1.21 [0.89 to 1.65] | 3.26 [2.02 to 5.28]
  4 weeks after 23-PPV: Serotype : 9V | 0.94 [0.71 to 1.24] | 3.84 [2.37 to 6.21]
  4 weeks after 23-PPV: Serotype : 10A | 1.14 [0.84 to 1.55] | 5.20 [3.27 to 8.28]
  4 weeks after 23-PPV: Serotype : 11F | 1.34 [1.03 to 1.74] | 4.74 [3.17 to 7.09]
  4 weeks after 23-PPV: Serotype : 12F | 1.13 [0.68 to 1.87] | 1.82 [1.11 to 2.99]
  4 weeks after 23-PPV: Serotype : 14 | 3.22 [2.29 to 4.54] | 12.51 [7.50 to 20.86]
  4 weeks after 23-PPV: Serotype : 15B | 1.57 [1.22 to 2.03] | 5.60 [3.20 to 9.80]
  4 weeks after 23-PPV: Serotype : 17F | 1.41 [1.09 to 1.84] | 5.33 [3.63 to 7.82]
  4 weeks after 23-PPV: Serotype : 18C | 1.55 [1.18 to 2.03] | 7.35 [4.39 to 12.31]
  4 weeks after 23-PPV: Serotype : 19A | 2.47 [1.71 to 3.55] | 8.96 [5.43 to 14.80]
  4 weeks after 23-PPV: Serotype : 19F | 1.57 [1.26 to 1.95] | 5.09 [3.25 to 7.97]
  4 weeks after 23-PPV: Serotype : 20 | 2.03 [1.52 to 2.71] | 3.74 [2.39 to 5.86]
  4 weeks after 23-PPV: Serotype : 22F | 1.10 [0.85 to 1.42] | 4.51 [2.93 to 6.95]
  4 weeks after 23-PPV: Serotype : 23F | 1.14 [0.90 to 1.46] | 2.90 [1.81 to 4.66]
  4 weeks after 23-PPV: Serotype : 33F | 1.44 [1.12 to 1.85] | 5.11 [3.25 to 8.05]

11. Secondary Outcome: Percentage of Participants With Positive Response Against Individual Pneumococcal Serotypes in 13-PCV
Description: as for outcome 8
Time Frame: 8 weeks after 23-PPV, which was 4 weeks after Group A1 participants received 13-PCV
Population: OC population included all randomized participants who completed the ISP.
Measure: Number; unit: percentage of participants
Arm/Group | Group A1 | Group A2 | Group B
Number analyzed (Participants) | 33 | 35 | 34
percentage of participants
  Serotype 1: number analyzed (Participants) | 31 | 34 | 34
  Serotype 1 | 54.8 | 38.2 | 100.0
  Serotype 2: number analyzed (Participants) | 31 | 34 | 34
  Serotype 2 | 54.8 | 44.1 | 97.1
  Serotype 3: number analyzed (Participants) | 31 | 34 | 34
  Serotype 3 | 35.5 | 29.4 | 85.3
  Serotype 4: number analyzed (Participants) | 31 | 34 | 34
  Serotype 4 | 32.3 | 23.5 | 88.2
  Serotype 5: number analyzed (Participants) | 31 | 34 | 34
  Serotype 5 | 38.7 | 44.1 | 97.1
  Serotype 6B: number analyzed (Participants) | 31 | 34 | 34
  Serotype 6B | 48.4 | 44.1 | 82.4
  Serotype 7F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 7F | 51.6 | 35.3 | 94.1
  Serotype 8: number analyzed (Participants) | 31 | 34 | 34
  Serotype 8 | 54.8 | 67.6 | 97.1
  Serotype 9N: number analyzed (Participants) | 31 | 34 | 34
  Serotype 9N | 45.2 | 47.1 | 82.4
  Serotype 9V: number analyzed (Participants) | 31 | 34 | 34
  Serotype 9V | 51.6 | 50.0 | 88.2
  Serotype 10A: number analyzed (Participants) | 31 | 34 | 34
  Serotype 10A | 29.0 | 29.4 | 91.2
  Serotype 11A: number analyzed (Participants) | 31 | 34 | 34
  Serotype 11A | 32.3 | 44.1 | 82.4
  Serotype 12F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 12F | 22.6 | 20.6 | 79.4
  Serotype 14: number analyzed (Participants) | 31 | 34 | 34
  Serotype 14 | 64.5 | 67.6 | 85.3
  Serotype 15B: number analyzed (Participants) | 31 | 34 | 34
  Serotype 15B | 35.5 | 38.2 | 88.2
  Serotype 17F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 17F | 41.9 | 44.1 | 88.2
  Serotype 18C: number analyzed (Participants) | 31 | 34 | 34
  Serotype 18C | 51.6 | 32.4 | 94.1
  Serotype 19A: number analyzed (Participants) | 31 | 34 | 34
  Serotype 19A | 58.1 | 35.3 | 88.2
  Serotype 19F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 19F | 41.9 | 29.4 | 88.2
  Serotype 20: number analyzed (Participants) | 31 | 34 | 34
  Serotype 20 | 25.8 | 14.7 | 85.3
  Serotype 22F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 22F | 38.7 | 23.5 | 91.2
  Serotype 23F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 23F | 48.4 | 29.4 | 76.5
  Serotype 33F: number analyzed (Participants) | 31 | 34 | 34
  Serotype 33F | 45.2 | 44.1 | 94.1
Statistical Analysis 1: Comparison: Group A1 vs Group B; Serotype 1- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -45.2, 95% CI 2-sided [-62.7 to -27.6]
Statistical Analysis 2: Comparison: Group A1 vs Group B; Serotype 2- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -42.2, 95% CI 2-sided [-60.6 to -23.8]
Statistical Analysis 3: Comparison: Group A1 vs Group B; Serotype 3- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -49.8, 95% CI 2-sided [-70.4 to -29.2]
Statistical Analysis 4: Comparison: Group A1 vs Group B; Serotype 4- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -56.0, 95% CI 2-sided [-75.7 to -36.3]
Statistical Analysis 5: Comparison: Group A1 vs Group B; Serotype 5- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -58.3, 95% CI 2-sided [-76.4 to -40.3]
Statistical Analysis 6: Comparison: Group A1 vs Group B; Serotype 6B- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -34.0, 95% CI 2-sided [-55.7 to -12.2]
Statistical Analysis 7: Comparison: Group A1 vs Group B; Serotype 7F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -42.5, 95% CI 2-sided [-61.8 to -23.2]
Statistical Analysis 8: Comparison: Group A1 vs Group B; Serotype 8- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -42.2, 95% CI 2-sided [-60.6 to -23.8]
Statistical Analysis 9: Comparison: Group A1 vs Group B; Serotype 9N- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -37.2, 95% CI 2-sided [-58.9 to -15.5]
Statistical Analysis 10: Comparison: Group A1 vs Group B; Serotype 9V- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -36.6, 95% CI 2-sided [-57.3 to -16.0]
Statistical Analysis 11: Comparison: Group A1 vs Group B; Serotype 10A- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -62.1, 95% CI 2-sided [-80.8 to -43.5]
Statistical Analysis 12: Comparison: Group A1 vs Group B; Serotype 11A- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -50.1, 95% CI 2-sided [-71.0 to -29.2]
Statistical Analysis 13: Comparison: Group A1 vs Group B; Serotype 12F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -56.8, 95% CI 2-sided [-76.9 to -36.8]
Statistical Analysis 14: Comparison: Group A1 vs Group B; Serotype 14- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -20.8, 95% CI 2-sided [-41.4 to -0.2]
Statistical Analysis 15: Comparison: Group A1 vs Group B; Serotype 15B- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -52.8, 95% CI 2-sided [-72.8 to -32.7]
Statistical Analysis 16: Comparison: Group A1 vs Group B; Serotype 17F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -46.3, 95% CI 2-sided [-66.8 to -25.8]
Statistical Analysis 17: Comparison: Group A1 vs Group B; Serotype 18C- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -42.5, 95% CI 2-sided [-61.8 to -23.2]
Statistical Analysis 18: Comparison: Group A1 vs Group B; Serotype 19A- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -30.2, 95% CI 2-sided [-50.6 to -9.7]
Statistical Analysis 19: Comparison: Group A1 vs Group B; Serotype 19F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -46.3, 95% CI 2-sided [-66.8 to -25.8]
Statistical Analysis 20: Comparison: Group A1 vs Group B; Serotype 20- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -59.5, 95% CI 2-sided [-79.0 to -40.0]
Statistical Analysis 21: Comparison: Group A1 vs Group B; Serotype 22F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -52.5, 95% CI 2-sided [-72.1 to -32.8]
Statistical Analysis 22: Comparison: Group A1 vs Group B; Serotype 23F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -28.1, 95% CI 2-sided [-50.7 to -5.4]
Statistical Analysis 23: Comparison: Group A1 vs Group B; Serotype 33F- Difference in positive response, Group A1 minus Group B; Test type: Superiority; Normal Distribution Approximation = -49.0, 95% CI 2-sided [-68.2 to -29.7]
Statistical Analysis 24: Comparison: Group A2 vs Group B; Serotype 1- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -61.8, 95% CI 2-sided [-78.1 to -45.4]
Statistical Analysis 25: Comparison: Group A2 vs Group B; Serotype 2- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -52.9, 95% CI 2-sided [-70.6 to -35.3]
Statistical Analysis 26: Comparison: Group A2 vs Group B; Serotype 3- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -55.9, 95% CI 2-sided [-75.3 to -36.5]
Statistical Analysis 27: Comparison: Group A2 vs Group B; Serotype 4- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -64.7, 95% CI 2-sided [-82.6 to -46.8]
Statistical Analysis 28: Comparison: Group A2 vs Group B; Serotype 5- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -52.9, 95% CI 2-sided [-70.6 to -35.3]
Statistical Analysis 29: Comparison: Group A2 vs Group B; Serotype 6B- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -38.2, 95% CI 2-sided [-59.3 to -17.2]
Statistical Analysis 30: Comparison: Group A2 vs Group B; Serotype 7F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -58.8, 95% CI 2-sided [-76.7 to -40.9]
Statistical Analysis 31: Comparison: Group A2 vs Group B; Serotype 8- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -29.4, 95% CI 2-sided [-46.1 to -12.7]
Statistical Analysis 32: Comparison: Group A2 vs Group B; Serotype 9N- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -35.3, 95% CI 2-sided [-56.4 to -14.2]
Statistical Analysis 33: Comparison: Group A2 vs Group B; Serotype 9V- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -38.2, 95% CI 2-sided [-58.2 to -18.2]
Statistical Analysis 34: Comparison: Group A2 vs Group B; Serotype 10A- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -61.8, 95% CI 2-sided [-79.8 to -43.7]
Statistical Analysis 35: Comparison: Group A2 vs Group B; Serotype 11A- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -38.2, 95% CI 2-sided [-59.3 to -17.2]
Statistical Analysis 36: Comparison: Group A2 vs Group B; Serotype 12F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -58.8, 95% CI 2-sided [-78.0 to -39.6]
Statistical Analysis 37: Comparison: Group A2 vs Group B; Serotype 14- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -17.6, 95% CI 2-sided [-37.4 to 2.1]
Statistical Analysis 38: Comparison: Group A2 vs Group B; Serotype 15B- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -50.0, 95% CI 2-sided [-69.6 to -30.4]
Statistical Analysis 39: Comparison: Group A2 vs Group B; Serotype 17F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -44.1, 95% CI 2-sided [-64.0 to -24.2]
Statistical Analysis 40: Comparison: Group A2 vs Group B; Serotype 18C- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -61.8, 95% CI 2-sided [-79.4 to -44.2]
Statistical Analysis 41: Comparison: Group A2 vs Group B; Serotype 19A- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -52.9, 95% CI 2-sided [-72.3 to -33.6]
Statistical Analysis 42: Comparison: Group A2 vs Group B; Serotype 19F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -58.8, 95% CI 2-sided [-77.6 to -40.1]
Statistical Analysis 43: Comparison: Group A2 vs Group B; Serotype 20- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -70.6, 95% CI 2-sided [-87.4 to -53.8]
Statistical Analysis 44: Comparison: Group A2 vs Group B; Serotype 22F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -67.6, 95% CI 2-sided [-84.8 to -50.5]
Statistical Analysis 45: Comparison: Group A2 vs Group B; Serotype 23F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -47.1, 95% CI 2-sided [-68.0 to -26.1]
Statistical Analysis 46: Comparison: Group A2 vs Group B; Serotype 33F- Difference in positive response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -50.0, 95% CI 2-sided [-68.5 to -31.5]

12. Secondary Outcome: Mean Level of Anti-Pneumococcal Antibody
Description: Serotype-specific antibody levels (IgG) were assessed by bead-based multi-analyte immunodetection (MAID).
Time Frame: Immediately prior to 23-PPV and 4 and 8 weeks after 23-PPV
Population: OC population included all randomized participants who completed the ISP.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group A1 | Group A2 | Group B
Number analyzed (Participants) | 33 | 35 | 34
mcg/mL
  Immediately prior to 23-PPV: Serotype : 1: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 1 | 0.84 [0.58 to 1.23] | 1.05 [0.68 to 1.62] | 1.02 [0.71 to 1.46]
  Immediately prior to 23-PPV: Serotype : 2: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 2 | 0.98 [0.63 to 1.52] | 1.27 [0.90 to 1.78] | 1.25 [0.93 to 1.69]
  Immediately prior to 23-PPV: Serotype : 3: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 3 | 0.93 [0.70 to 1.23] | 1.35 [0.75 to 2.42] | 0.95 [0.66 to 1.36]
  Immediately prior to 23-PPV: Serotype : 4: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 4 | 0.37 [0.29 to 0.47] | 0.88 [0.46 to 1.66] | 0.59 [0.40 to 0.88]
  Immediately prior to 23-PPV: Serotype : 5: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 5 | 0.77 [0.57 to 1.05] | 1.22 [0.76 to 1.97] | 1.31 [0.91 to 1.89]
  Immediately prior to 23-PPV: Serotype : 6B: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 6B | 0.64 [0.46 to 0.88] | 1.08 [0.70 to 1.68] | 0.92 [0.60 to 1.39]
  Immediately prior to 23-PPV: Serotype : 7F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 7F | 1.04 [0.77 to 1.40] | 0.76 [0.57 to 1.00] | 0.94 [0.70 to 1.27]
  Immediately prior to 23-PPV: Serotype : 8: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 8 | 0.89 [0.62 to 1.27] | 0.96 [0.58 to 1.57] | 0.91 [0.59 to 1.38]
  Immediately prior to 23-PPV: Serotype : 9N: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 9N | 0.59 [0.40 to 0.86] | 0.98 [0.62 to 1.54] | 1.06 [0.68 to 1.64]
  Immediately prior to 23-PPV: Serotype : 9V: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 9V | 0.51 [0.40 to 0.65] | 1.09 [0.63 to 1.90] | 0.74 [0.50 to 1.11]
  Immediately prior to 23-PPV: Serotype : 10A: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 10A | 0.73 [0.52 to 1.03] | 1.01 [0.67 to 1.53] | 0.96 [0.73 to 1.26]
  Immediately prior to 23-PPV: Serotype : 11F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 11F | 1.09 [0.75 to 1.58] | 1.08 [0.69 to 1.71] | 1.03 [0.69 to 1.52]
  Immediately prior to 23-PPV: Serotype : 12F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 12F | 0.67 [0.49 to 0.93] | 0.89 [0.35 to 2.24] | 0.54 [0.35 to 0.83]
  Immediately prior to 23-PPV: Serotype : 14: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 14 | 0.98 [0.68 to 1.42] | 1.67 [1.04 to 2.69] | 1.09 [0.71 to 1.68]
  Immediately prior to 23-PPV: Serotype : 15B: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 15B | 0.68 [0.50 to 0.91] | 0.96 [0.76 to 1.23] | 1.18 [0.73 to 1.92]
  Immediately prior to 23-PPV: Serotype : 17F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 17F | 0.84 [0.58 to 1.22] | 0.94 [0.68 to 1.30] | 1.05 [0.75 to 1.48]
  Immediately prior to 23-PPV: Serotype : 18C: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 18C | 1.11 [0.73 to 1.70] | 1.04 [0.75 to 1.46] | 1.14 [0.79 to 1.64]
  Immediately prior to 23-PPV: Serotype : 19A: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 19A | 1.24 [0.88 to 1.74] | 1.99 [1.15 to 3.43] | 2.09 [1.26 to 3.46]
  Immediately prior to 23-PPV: Serotype : 19F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 19F | 1.06 [0.80 to 1.41] | 1.13 [0.83 to 1.53] | 1.16 [0.80 to 1.67]
  Immediately prior to 23-PPV: Serotype : 20: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 20 | 1.38 [0.93 to 2.06] | 2.13 [1.39 to 3.25] | 1.29 [0.89 to 1.87]
  Immediately prior to 23-PPV: Serotype : 22F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 22F | 0.58 [0.43 to 0.78] | 0.98 [0.60 to 1.59] | 0.82 [0.55 to 1.20]
  Immediately prior to 23-PPV: Serotype : 23F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 23F | 0.68 [0.51 to 0.91] | 0.77 [0.50 to 1.20] | 0.96 [0.66 to 1.41]
  Immediately prior to 23-PPV: Serotype : 33F: number analyzed (Participants) | 33 | 34 | 34
  Immediately prior to 23-PPV: Serotype : 33F | 0.87 [0.62 to 1.22] | 1.05 [0.75 to 1.46] | 0.67 [0.52 to 0.85]
  4 weeks after 23-PPV: Serotype : 1 | 1.16 [0.83 to 1.62] | 1.46 [1.04 to 2.06] | 11.58 [7.72 to 17.38]
  4 weeks after 23-PPV: Serotype : 2 | 1.78 [1.23 to 2.57] | 1.79 [1.26 to 2.56] | 9.41 [6.80 to 13.01]
  4 weeks after 23-PPV: Serotype : 3 | 1.58 [1.12 to 2.23] | 1.56 [1.03 to 2.38] | 2.76 [1.72 to 4.42]
  4 weeks after 23-PPV: Serotype : 4 | 1.15 [0.59 to 2.24] | 1.90 [1.11 to 3.23] | 2.02 [1.32 to 3.08]
  4 weeks after 23-PPV: Serotype : 5 | 1.09 [0.78 to 1.51] | 1.44 [0.97 to 2.13] | 10.16 [5.69 to 18.15]
  4 weeks after 23-PPV: Serotype : 6B | 1.28 [0.78 to 2.10] | 1.69 [1.02 to 2.81] | 3.94 [2.12 to 7.33]
  4 weeks after 23-PPV: Serotype : 7F | 1.73 [1.17 to 2.56] | 1.10 [0.82 to 1.47] | 4.92 [2.99 to 8.09]
  4 weeks after 23-PPV: Serotype : 8 | 1.59 [1.10 to 2.29] | 1.97 [1.30 to 2.99] | 9.04 [6.42 to 12.73]
  4 weeks after 23-PPV: Serotype : 9N | 1.08 [0.71 to 1.63] | 1.35 [0.86 to 2.12] | 3.26 [2.02 to 5.28]
  4 weeks after 23-PPV: Serotype : 9V | 0.68 [0.50 to 0.93] | 1.21 [0.80 to 1.82] | 3.84 [2.37 to 6.21]
  4 weeks after 23-PPV: Serotype : 10A | 0.84 [0.56 to 1.25] | 1.49 [0.95 to 2.32] | 5.20 [3.27 to 8.28]
  4 weeks after 23-PPV: Serotype : 11F | 1.43 [1.02 to 2.03] | 1.27 [0.86 to 1.87] | 4.74 [3.17 to 7.09]
  4 weeks after 23-PPV: Serotype : 12F | 0.71 [0.40 to 1.25] | 1.66 [0.78 to 3.52] | 1.82 [1.11 to 2.99]
  4 weeks after 23-PPV: Serotype : 14 | 2.02 [1.32 to 3.09] | 4.83 [2.97 to 7.86] | 12.51 [7.50 to 20.86]
  4 weeks after 23-PPV: Serotype : 15B | 1.24 [0.81 to 1.92] | 1.91 [1.43 to 2.55] | 5.60 [3.20 to 9.80]
  4 weeks after 23-PPV: Serotype : 17F | 1.51 [0.98 to 2.32] | 1.35 [0.97 to 1.89] | 5.33 [3.63 to 7.82]
  4 weeks after 23-PPV: Serotype : 18C | 2.05 [1.37 to 3.08] | 1.19 [0.84 to 1.67] | 7.35 [4.39 to 12.31]
  4 weeks after 23-PPV: Serotype : 19A | 2.04 [1.35 to 3.07] | 2.95 [1.64 to 5.33] | 8.96 [5.43 to 14.80]
  4 weeks after 23-PPV: Serotype : 19F | 1.56 [1.20 to 2.03] | 1.58 [1.11 to 2.25] | 5.09 [3.25 to 7.97]
  4 weeks after 23-PPV: Serotype : 20 | 1.63 [1.14 to 2.33] | 2.50 [1.61 to 3.87] | 3.74 [2.39 to 5.86]
  4 weeks after 23-PPV: Serotype : 22F | 1.06 [0.71 to 1.58] | 1.14 [0.83 to 1.57] | 4.51 [2.93 to 6.95]
  4 weeks after 23-PPV: Serotype : 23F | 1.11 [0.77 to 1.60] | 1.18 [0.86 to 1.62] | 2.90 [1.81 to 4.66]
  4 weeks after 23-PPV: Serotype : 33F | 1.14 [0.82 to 1.58] | 1.82 [1.27 to 2.62] | 5.11 [3.25 to 8.05]
  8 weeks after 23-PPV: Serotype : 1: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 1 | 1.32 [0.92 to 1.91] | 1.34 [0.96 to 1.86] | 11.38 [7.66 to 16.92]
  8 weeks after 23-PPV: Serotype : 2: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 2 | 1.86 [1.16 to 2.99] | 1.67 [1.19 to 2.36] | 10.07 [7.33 to 13.83]
  8 weeks after 23-PPV: Serotype : 3: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 3 | 1.68 [1.13 to 2.51] | 1.33 [0.89 to 2.00] | 2.99 [1.89 to 4.73]
  8 weeks after 23-PPV: Serotype : 4: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 4 | 1.36 [0.64 to 2.89] | 1.84 [1.07 to 3.16] | 1.96 [1.30 to 2.96]
  8 weeks after 23-PPV: Serotype : 5: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 5 | 1.18 [0.85 to 1.64] | 1.21 [0.83 to 1.74] | 9.17 [5.06 to 16.60]
  8 weeks after 23-PPV: Serotype : 6B: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 6B | 1.72 [0.98 to 3.01] | 1.94 [1.18 to 3.19] | 4.85 [2.58 to 9.10]
  8 weeks after 23-PPV: Serotype : 7F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 7F | 1.73 [1.23 to 2.43] | 1.07 [0.78 to 1.46] | 4.95 [3.02 to 8.10]
  8 weeks after 23-PPV: Serotype : 8: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 8 | 1.83 [1.24 to 2.71] | 1.80 [1.22 to 2.65] | 8.57 [6.03 to 12.19]
  8 weeks after 23-PPV: Serotype : 9N: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 9N | 1.09 [0.75 to 1.60] | 1.10 [0.74 to 1.63] | 3.37 [2.11 to 5.40]
  8 weeks after 23-PPV: Serotype : 9V: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 9V | 0.88 [0.65 to 1.18] | 1.08 [0.73 to 1.58] | 4.44 [2.75 to 7.16]
  8 weeks after 23-PPV: Serotype : 10A: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 10A | 1.05 [0.58 to 1.88] | 1.38 [0.91 to 2.12] | 5.75 [3.63 to 9.11]
  8 weeks after 23-PPV: Serotype : 11F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 11F | 1.29 [0.91 to 1.84] | 1.08 [0.74 to 1.57] | 4.42 [2.95 to 6.61]
  8 weeks after 23-PPV: Serotype : 12F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 12F | 0.91 [0.57 to 1.43] | 2.33 [1.09 to 4.98] | 2.13 [1.30 to 3.49]
  8 weeks after 23-PPV: Serotype : 14: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 14 | 2.06 [1.38 to 3.08] | 4.87 [3.05 to 7.79] | 12.29 [7.38 to 20.47]
  8 weeks after 23-PPV: Serotype : 15B: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 15B | 1.25 [0.80 to 1.94] | 1.66 [1.24 to 2.22] | 5.76 [3.34 to 9.92]
  8 weeks after 23-PPV: Serotype : 17F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 17F | 1.48 [0.88 to 2.46] | 1.29 [0.98 to 1.71] | 5.57 [3.76 to 8.25]
  8 weeks after 23-PPV: Serotype : 18C: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 18C | 2.29 [1.54 to 3.40] | 1.18 [0.85 to 1.62] | 7.14 [4.37 to 11.65]
  8 weeks after 23-PPV: Serotype : 19A: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 19A | 2.35 [1.53 to 3.59] | 3.21 [1.76 to 5.84] | 9.56 [5.87 to 15.56]
  8 weeks after 23-PPV: Serotype : 19F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 19F | 1.74 [1.30 to 2.33] | 1.56 [1.09 to 2.24] | 4.91 [3.12 to 7.73]
  8 weeks after 23-PPV: Serotype : 20: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 20 | 1.73 [1.13 to 2.66] | 2.59 [1.71 to 3.92] | 3.56 [2.31 to 5.50]
  8 weeks after 23-PPV: Serotype : 22F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 22F | 1.22 [0.70 to 2.12] | 1.09 [0.79 to 1.50] | 4.69 [3.11 to 7.09]
  8 weeks after 23-PPV: Serotype : 23F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 23F | 1.21 [0.83 to 1.77] | 1.07 [0.79 to 1.44] | 2.44 [1.58 to 3.76]
  8 weeks after 23-PPV: Serotype : 33F: number analyzed (Participants) | 31 | 35 | 34
  8 weeks after 23-PPV: Serotype : 33F | 1.36 [0.96 to 1.92] | 1.68 [1.23 to 2.30] | 5.01 [3.16 to 7.95]

13. Secondary Outcome: Percentage of Participants With Seroprotection
Description: Seroprotection was defined as specific hemagglutination inhibition (HI) titers >40 at 4 weeks after vaccination.
Time Frame: 4 weeks after seasonal influenza vaccine administration
Population: OC population included all randomized participants who completed the ISP. Analysis applies to participants who received influenza vaccine (Groups A2 and B).
Measure: Number; unit: percentage of participants
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
percentage of participants
  Strain = H1N1CA09: number analyzed (Participants) | 35 | 33
  Strain = H1N1CA09 | 71.4 | 97.0
  Strain = BPHU13: number analyzed (Participants) | 33 | 31
  Strain = BPHU13 | 66.7 | 80.6
  Strain = H3N2SW13: number analyzed (Participants) | 30 | 27
  Strain = H3N2SW13 | 66.7 | 92.6
  Strain = BBRIS08: number analyzed (Participants) | 18 | 16
  Strain = BBRIS08 | 55.6 | 75.0
  Strain = AHK4801: number analyzed (Participants) | 5 | 6
  Strain = AHK4801 | 80.0 | 83.3
Statistical Analysis 1: Comparison: Group A2 vs Group B; Strain = H1N1CA09 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -25.5, 95% CI 2-sided [-41.6 to -9.5]
Statistical Analysis 2: Comparison: Group A2 vs Group B; Strain = BPHU13 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -14.0, 95% CI 2-sided [-35.2 to 7.3]
Statistical Analysis 3: Comparison: Group A2 vs Group B; Strain = H3N2SW13 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -25.9, 95% CI 2-sided [-45.5 to -6.4]
Statistical Analysis 4: Comparison: Group A2 vs Group B; Strain = BBRIS08 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -19.4, 95% CI 2-sided [-50.7 to 11.8]
Statistical Analysis 5: Comparison: Group A2 vs Group B; Strain = AHK4801 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -3.3, 95% CI 2-sided [-49.4 to 42.7]

14. Secondary Outcome: Percentage of Participants With 2-Fold Increase in Strain-Specific HI Titers
Description: 2-fold increase from prevaccination HI titer.
Time Frame: 4 weeks after seasonal influenza vaccine administration
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
percentage of participants
  Strain = H1N1CA09: number analyzed (Participants) | 35 | 32
  Strain = H1N1CA09 | 45.7 | 87.5
  Strain = BPHU13: number analyzed (Participants) | 33 | 30
  Strain = BPHU13 | 42.4 | 80.0
  Strain = H3N2SW13: number analyzed (Participants) | 30 | 26
  Strain = H3N2SW13 | 36.7 | 96.2
  Strain = BBRIS08: number analyzed (Participants) | 18 | 15
  Strain = BBRIS08 | 27.8 | 73.3
  Strain = AHK4801: number analyzed (Participants) | 5 | 6
  Strain = AHK4801 | 80.0 | 83.3
Statistical Analysis 1: Comparison: Group A2 vs Group B; Strain = H1N1CA09 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -41.8, 95% CI 2-sided [-61.9 to -21.7]
Statistical Analysis 2: Comparison: Group A2 vs Group B; Strain = BPHU13 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -37.6, 95% CI 2-sided [-59.7 to -15.5]
Statistical Analysis 3: Comparison: Group A2 vs Group B; Strain = H3N2SW13 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -59.5, 95% CI 2-sided [-78.2 to -40.7]
Statistical Analysis 4: Comparison: Group A2 vs Group B; Strain = BBRIS08 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -45.6, 95% CI 2-sided [-76.0 to -15.1]
Statistical Analysis 5: Comparison: Group A2 vs Group B; Strain = AHK4801 (Group A2 minus Group B); Test type: Superiority; Normal Distribution Approximation = -3.3, 95% CI 2-sided [-49.4 to 42.7]

15. Secondary Outcome: Percentage of Participants With 4-Fold Increase in Strain-Specific HI Titers
Description: 4-fold increase from prevaccination HI titer.
Time Frame: 4 weeks after seasonal influenza vaccine administration
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
percentage of participants
  Strain = H1N1CA09: number analyzed (Participants) | 35 | 32
  Strain = H1N1CA09 | 20.0 | 81.3
  Strain = BPHU13: number analyzed (Participants) | 33 | 30
  Strain = BPHU13 | 15.2 | 70.0
  Strain = H3N2SW13: number analyzed (Participants) | 30 | 26
  Strain = H3N2SW13 | 10.0 | 92.3
  Strain = BBRIS08: number analyzed (Participants) | 18 | 15
  Strain = BBRIS08 | 16.7 | 53.3
  Strain = AHK4801: number analyzed (Participants) | 5 | 6
  Strain = AHK4801 | 60.0 | 66.7
Statistical Analysis 1: Comparison: Group A2 vs Group B; Strain = H1N1CA09 - Difference in at least 4-fold response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -61.3, 95% CI 2-sided [-80.2 to -42.3]
Statistical Analysis 2: Comparison: Group A2 vs Group B; Strain = BPHU13 - Difference in at least 4-fold response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -54.8, 95% CI 2-sided [-75.3 to -34.4]
Statistical Analysis 3: Comparison: Group A2 vs Group B; Strain = H3N2SW13 - Difference in at least 4-fold response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -82.3, 95% CI 2-sided [-97.1 to -67.5]
Statistical Analysis 4: Comparison: Group A2 vs Group B; Strain = BBRIS08 - Difference in at least 4-fold response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -36.7, 95% CI 2-sided [-67.2 to -6.1]
Statistical Analysis 5: Comparison: Group A2 vs Group B; Strain = AHK4801 - Difference in at least 4-fold response, Group A2 minus Group B; Test type: Superiority; Normal Distribution Approximation = -6.7, 95% CI 2-sided [-63.8 to 50.5]

16. Secondary Outcome: Percentage of Participants With Seroconversion
Description: Seroconversion at 4 weeks after vaccination defined, as per protocol, as a prevaccination HI titer <10 and an HI titer >40 at 4 weeks after vaccination. Seroconversion at 4 weeks after vaccination, defined per FDA guidance, as either a) a pre-vaccination HI titer <10 and HI titer >/= 40 at 4 weeks after vaccination, or b) a pre-vaccination HI titer >/= 10 and at least 4-fold increase in HI antibody titer at 4 weeks after vaccination.
Time Frame: 4 weeks after influenza immunization
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
percentage of participants
  Strain = H1N1CA09 (as per FDA guidance): number analyzed (Participants) | 35 | 32
  Strain = H1N1CA09 (as per FDA guidance) | 20.0 | 81.3
  Strain = H1N1CA09 (as per protocol): number analyzed (Participants) | 7 | 9
  Strain = H1N1CA09 (as per protocol) | 42.9 | 88.9
  Strain = BPHU13 (as per FDA guidance): number analyzed (Participants) | 33 | 30
  Strain = BPHU13 (as per FDA guidance) | 12.1 | 70.0
  Strain = BPHU13 (as per protocol): number analyzed (Participants) | 4 | 9
  Strain = BPHU13 (as per protocol) | 0 | 55.6
  Strain = H3N2SW13 (as per FDA guidance): number analyzed (Participants) | 30 | 26
  Strain = H3N2SW13 (as per FDA guidance) | 10.0 | 88.5
  Strain = H3N2SW13 (as per protocol): number analyzed (Participants) | 5 | 9
  Strain = H3N2SW13 (as per protocol) | 20.0 | 77.8
  Strain = BBRIS08 (as per FDA guidance): number analyzed (Participants) | 18 | 15
  Strain = BBRIS08 (as per FDA guidance) | 16.7 | 53.3
  Strain = BBRIS08 (as per protocol): number analyzed (Participants) | 3 | 4
  Strain = BBRIS08 (as per protocol) | 0 | 25.0
  Strain = AHK4801 (as per FDA guidance): number analyzed (Participants) | 5 | 6
  Strain = AHK4801 (as per FDA guidance) | 60.0 | 66.7
  Strain = AHK4801 (as per protocol): number analyzed (Participants) | 0 | 2
  Strain = AHK4801 (as per protocol) |  | 100.0
Statistical Analysis 1: Comparison: Group A2 vs Group B; Strain = H1N1CA09 (Group A2 minus Group B) [FDA]; Test type: Superiority; Normal Distribution Approximation = -61.3, 95% CI 2-sided [-80.2 to -42.3]
Statistical Analysis 2: Comparison: Group A2 vs Group B; Strain = H1N1CA09 (Group A2 minus Group B) [Protocol]; Test type: Superiority; Normal Distribution Approximation = -46.0, 95% CI 2-sided [-88.0 to -4.0]
Statistical Analysis 3: Comparison: Group A2 vs Group B; Strain = BPHU13 (Group A2 minus Group B) [FDA]; Test type: Superiority; Normal Distribution Approximation = -57.9, 95% CI 2-sided [-77.7 to -38.1]
Statistical Analysis 4: Comparison: Group A2 vs Group B; Strain = BPHU13 (Group A2 minus Group B) [Protocol]; Test type: Superiority; Normal Distribution Approximation = -55.6, 95% CI 2-sided [-88.0 to -23.1]
Statistical Analysis 5: Comparison: Group A2 vs Group B; Strain = H3N2SW13 (Group A2 minus Group B) [FDA]; Test type: Superiority; Normal Distribution Approximation = -78.5, 95% CI 2-sided [-94.8 to -62.2]
Statistical Analysis 6: Comparison: Group A2 vs Group B; Strain = H3N2SW13 (Group A2 minus Group B) [Protocol]; Test type: Superiority; Normal Distribution Approximation = -57.8, 95% CI 2-sided [-100.0 to -13.4]
Statistical Analysis 7: Comparison: Group A2 vs Group B; Strain = BBRIS08 (Group A2 minus Group B) [FDA]; Test type: Superiority; Normal Distribution Approximation = -36.7, 95% CI 2-sided [-67.2 to -6.1]
Statistical Analysis 8: Comparison: Group A2 vs Group B; Strain = BBRIS08 (Group A2 minus Group B) [Protocol]; Test type: Superiority; Normal Distribution Approximation = -25.0, 95% CI 2-sided [-67.4 to 17.4]
Statistical Analysis 9: Comparison: Group A2 vs Group B; Strain = AHK4801 (Group A2 minus Group B) [FDA]; Test type: Superiority; Normal Distribution Approximation = -6.7, 95% CI 2-sided [-63.8 to 50.5]

17. Secondary Outcome: Strain-Specific Geometric Mean Titer Levels
Description: Geometric mean titers (GMTs) in participants in Groups A2 and B were measured 4 weeks after vaccination.
Time Frame: Baseline and Week 4
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: hemagglutination inhibition titers
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
hemagglutination inhibition titers
  Prior to influenza vaccine: Strain = H1N1CA09: number analyzed (Participants) | 28 | 24
  Prior to influenza vaccine: Strain = H1N1CA09 | 126.5 [78.2 to 204.4] | 86.0 [55.4 to 133.6]
  4 weeks after influenza vaccine: Strain = H1N1CA09: number analyzed (Participants) | 32 | 33
  4 weeks after influenza vaccine: Strain = H1N1CA09 | 154.8 [103.8 to 230.8] | 390.8 [264.0 to 578.4]
  Prior to influenza vaccine: Strain = BPHU13: number analyzed (Participants) | 29 | 22
  Prior to influenza vaccine: Strain = BPHU13 | 67.7 [49.5 to 92.4] | 54.0 [34.6 to 84.3]
  4 weeks after influenza vaccine: Strain = BPHU13: number analyzed (Participants) | 31 | 29
  4 weeks after influenza vaccine: Strain = BPHU13 | 84.6 [64.3 to 111.3] | 243.1 [156.3 to 377.9]
  Prior to influenza vaccine: Strain = H3N2SW13: number analyzed (Participants) | 25 | 17
  Prior to influenza vaccine: Strain = H3N2SW13 | 110.0 [72.9 to 166.0] | 62.6 [41.2 to 95.2]
  4 weeks after influenza vaccine: Strain = H3N2SW13: number analyzed (Participants) | 26 | 25
  4 weeks after influenza vaccine: Strain = H3N2SW13 | 134.5 [94.9 to 190.5] | 342.8 [219.1 to 536.3]
  Prior to influenza vaccine: Strain = BBRIS08: number analyzed (Participants) | 15 | 12
  Prior to influenza vaccine: Strain = BBRIS08 | 49.3 [35.2 to 69.0] | 71.3 [35.7 to 142.3]
  4 weeks after influenza vaccine: Strain = BBRIS08: number analyzed (Participants) | 16 | 13
  4 weeks after influenza vaccine: Strain = BBRIS08 | 65.8 [43.6 to 99.3] | 311.7 [167.4 to 580.5]
  Prior to influenza vaccine: Strain = AHK4801: number analyzed (Participants) | 5 | 5
  Prior to influenza vaccine: Strain = AHK4801 | 52.8 [21.0 to 132.6] | 45.9 [32.4 to 65.2]
  4 weeks after influenza vaccine: Strain = AHK4801: number analyzed (Participants) | 5 | 6
  4 weeks after influenza vaccine: Strain = AHK4801 | 121.3 [70.4 to 208.8] | 127.0 [55.1 to 292.7]

18. Secondary Outcome: Ratio of Strain-Specific Geometric Mean Titer Levels Postvaccination to Prevaccination
Description: Strain-specific GMT ratios were calculated as post-vaccination : pre-vaccination.
Time Frame: Immediately prior to and 4 weeks after influenza vaccine
Population: as for outcome 13
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Group A2 | Group B
Number analyzed (Participants) | 35 | 34
ratio
  Strain = H1N1CA09: number analyzed (Participants) | 28 | 23
  Strain = H1N1CA09 | 1.31 (1.04) | 5.74 (21.05)
  Strain = BPHU13: number analyzed (Participants) | 29 | 21
  Strain = BPHU13 | 1.35 (1.62) | 6.45 (28.31)
  Strain = H3N2SW13: number analyzed (Participants) | 25 | 16
  Strain = H3N2SW13 | 1.25 (0.94) | 8.18 (11.70)
  Strain = BBRIS08: number analyzed (Participants) | 15 | 11
  Strain = BBRIS08 | 1.38 (1.90) | 4.68 (9.19)
  Strain = AHK4801: number analyzed (Participants) | 5 | 4
  Strain = AHK4801 | 2.30 (1.60) | 2.83 (3.34)

19. Secondary Outcome: Magnetic Resonance Imaging (MRI) Parameters: Volume of T2 Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: cubic centimeters (cm^3)
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
cubic centimeters (cm^3) | 10.76 (13.31) | 7.53 (8.20)

20. Secondary Outcome: MRI Parameters: Number of T2 Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
lesions | 57.94 (45.43) | 45.53 (28.61)

21. Secondary Outcome: MRI Parameters: Categorical Number of T2 Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP. Data are reported for evaluable participants.
Measure: Number; unit: participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
participants
  Baseline: 0-5 lesions: number analyzed (Participants) | 66 | 34
  Baseline: 0-5 lesions | 1 | 0
  Baseline: 6-9 lesions: number analyzed (Participants) | 66 | 34
  Baseline: 6-9 lesions | 1 | 1
  Baseline: >9 lesions: number analyzed (Participants) | 66 | 34
  Baseline: >9 lesions | 64 | 33

22. Secondary Outcome: MRI Parameters: Number of Gadolinium (Gd)-Enhancing T1 Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
lesions | 2.85 (10.93) | 0.62 (2.65)

23. Secondary Outcome: MRI Parameters: Categorical Number of Gd-enhancing T1 Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP. Data are reported for evaluable participants.
Measure: Number; unit: participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
participants
  Baseline: 0 lesions: number analyzed (Participants) | 65 | 34
  Baseline: 0 lesions | 44 | 31
  Baseline: 1 lesions: number analyzed (Participants) | 65 | 34
  Baseline: 1 lesions | 8 | 0
  Baseline: 2 lesions: number analyzed (Participants) | 65 | 34
  Baseline: 2 lesions | 2 | 1
  Baseline: 3 lesions: number analyzed (Participants) | 65 | 34
  Baseline: 3 lesions | 2 | 0
  Baseline: >=4 lesions: number analyzed (Participants) | 65 | 34
  Baseline: >=4 lesions | 9 | 2

24. Secondary Outcome: MRI Parameters: Normalized Brain Volume
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
cm^3 | 1470.51 (77.83) | 1456.35 (70.03)

25. Secondary Outcome: MRI Parameters: Volume of T2 Lesions: White Matter Volume
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
cm^3 | 808.22 (60.11) | 794.53 (47.58)

26. Secondary Outcome: MRI Parameters: Cortical Grey Matter Volume
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
cm^3 | 521.19 (35.28) | 519.70 (36.18)

27. Secondary Outcome: MRI Parameters: T1 Unenhancing Lesion Volume
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
cm^3 | 1.85 (2.75) | 1.31 (1.75)

28. Secondary Outcome: MRI Parameters: Total Number of Lesions
Description: MRI assessments done to evaluate the long-term effects of ocrelizumab on MRI parameters.
Time Frame: Baseline
Population: OC population included all randomized participants who completed the ISP.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
lesions | 25.51 (27.76) | 18.85 (15.99)

29. Secondary Outcome: Cellular Immune Response Assessed by Flow Cytometry
Description: Flow cytometry is a laser-based technology commonly used for cell counting and sorting. In this study, this outcome measure is focusing on a single variable, CD19 count (total B cells). LLN = 80 cells/ul.
  Repleted is defined as CD19 >= LLN or baseline, whichever is lower.
Time Frame: Days 1, 15, 85, 112, 140 and 169
Population: Safety population included all participants who received any ocrelizumab or any vaccine. Data are reported for evaluable participants.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants
  >=lower limit of normal range (LLN) - Day 1: number analyzed (Participants) | 67 | 33
  >=lower limit of normal range (LLN) - Day 1 | 97.0 | 97.0
  <LLN - Day 1: number analyzed (Participants) | 67 | 34
  <LLN - Day 1 | 3.0 | 3.0
  CD19 repleted - Day 1: number analyzed (Participants) | 67 | 34
  CD19 repleted - Day 1 | 100.0 | 100.0
  CD19 not repleted - Day 1: number analyzed (Participants) | 67 | 34
  CD19 not repleted - Day 1 | 0 | 0
  >=LLN - Day 15: number analyzed (Participants) | 66 | 0
  >=LLN - Day 15 | 0 |
  <LLN - Day 15: number analyzed (Participants) | 66 | 0
  <LLN - Day 15 | 100.0 |
  CD19 repleted - Day 15: number analyzed (Participants) | 66 | 0
  CD19 repleted - Day 15 | 0 |
  CD19 not repleted - Day 15: number analyzed (Participants) | 66 | 0
  CD19 not repleted - Day 15 | 100.0 |
  >=LLN - Day 85: number analyzed (Participants) | 63 | 32
  >=LLN - Day 85 | 0 | 90.6
  <LLN - Day 85: number analyzed (Participants) | 63 | 32
  <LLN - Day 85 | 100.0 | 9.4
  CD19 repleted - Day 85: number analyzed (Participants) | 63 | 32
  CD19 repleted - Day 85 | 0 | 90.6
  CD19 not repleted - Day 85: number analyzed (Participants) | 63 | 32
  CD19 not repleted - Day 85 | 100.0 | 9.4
  >=LLN - Day 112: number analyzed (Participants) | 64 | 0
  >=LLN - Day 112 | 0 |
  <LLN - Day 112: number analyzed (Participants) | 64 | 0
  <LLN - Day 112 | 100.0 |
  CD19 repleted - Day 112: number analyzed (Participants) | 64 | 0
  CD19 repleted - Day 112 | 0 |
  CD19 not repleted - Day 112: number analyzed (Participants) | 64 | 0
  CD19 not repleted - Day 112 | 100.0 |
  >=LLN - Day 140: number analyzed (Participants) | 67 | 0
  >=LLN - Day 140 | 1.5 |
  <LLN - Day 140: number analyzed (Participants) | 67 | 0
  <LLN - Day 140 | 98.5 |
  CD19 repleted - Day 140: number analyzed (Participants) | 67 | 0
  CD19 repleted - Day 140 | 1.5 |
  CD19 not repleted - Day 140: number analyzed (Participants) | 67 | 0
  CD19 not repleted - Day 140 | 98.5 |
  >=LLN - Day 169: number analyzed (Participants) | 64 | 0
  >=LLN - Day 169 | 3.1 |
  <LLN - Day 169: number analyzed (Participants) | 64 | 0
  <LLN - Day 169 | 96.9 |
  CD19 repleted - Day 169: number analyzed (Participants) | 64 | 0
  CD19 repleted - Day 169 | 3.1 |
  CD19 not repleted - Day 169: number analyzed (Participants) | 64 | 0
  CD19 not repleted - Day 169 | 96.9 |

30. Secondary Outcome: Total Immunoglobulin
Time Frame: Days 1, 85, and 169
Population: Safety population included all participants who received any ocrelizumab or any vaccine.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
grams per liter (g/L)
  Day 1 | 13.45 (2.75) | 14.05 (3.01)
  Day 85 | 13.45 (2.80) | 14.53 (3.19)
  Day 169: number analyzed (Participants) | 67 | 0
  Day 169 | 13.26 (2.62) |

31. Secondary Outcome: Percentage of Participants With Anti-Drug Antibody Formation
Description: Anti-Drug Antibodies (ADA) may induce unwanted side effects, especially in biotechnology-derived pharmaceuticals, such as therapeutic antibodies and growth factors.
Time Frame: Up to 24 Weeks (ISP)
Population: Safety population included all participants who received any ocrelizumab or any vaccine. Data are reported for participants with measurable ADA samples.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants
  Baseline: number analyzed (Participants) | 68 | 0
  Baseline | 0 |
  Post-baseline: number analyzed (Participants) | 68 | 26
  Post-baseline | 0 | 0

32. Secondary Outcome: Percentage of Participants With Adverse Events (AEs), Serious AEs, or AEs Leading to Study Discontinuation
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious AE is any AE that is fatal, life-threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug, or is a significant medical event in the investigator's judgment.
Time Frame: During ISP (24 weeks for Group A and 12 weeks for Group B)
Population: Safety population included all participants who received any ocrelizumab or any vaccine.
Measure: Number; unit: percentage of participants
Arm/Group | Group A (A1 + A2) | Group B
Number analyzed (Participants) | 68 | 34
percentage of participants
  AEs | 82.4 | 50.0
  Serious AEs | 0 | 0
  AEs Leading to Study Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up 5 years, 10 months, 26 days
Description: Group A received 600 mg OCR and then vaccine challenge Group B received no OCR, just vaccine challenge.
Groups:
- Group B: Participants received immunizations (TT-containing adsorbed vaccine, 23-PPV, influenza vaccine, and repeated administration with KLH) on Day 1 until Week 12 of the immunization period. No study drug was administered.
Arm/Group | Group A1 | Group A2 | Group B
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 5/33 | 5/35 | 6/34
Other Adverse Events (participants affected / at risk) | 31/33 | 34/35 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A1 (N=33) | Group A2 (N=35) | Group B (N=34)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER DISSEMINATED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
HEAD INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SARS-COV-2 TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 1 (1)
LOBULAR BREAST CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
CAROTID ARTERY ANEURYSM (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A1 (N=33) | Group A2 (N=35) | Group B (N=34)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2)
PALPITATIONS (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 4 (4) | 2 (2) | 1 (1)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
VISION BLURRED (Eye disorders) | 6 (7) | 1 (1) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
ANAL INCONTINENCE (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 6 (7) | 5 (5) | 3 (4)
DYSPEPSIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (8) | 8 (11) | 5 (6)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (4) | 2 (2) | 4 (4)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 1 (1)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2) | 0 (0)
CYST (General disorders) | 0 (0) | 2 (2) | 0 (0)
FATIGUE (General disorders) | 16 (23) | 10 (13) | 7 (7)
GAIT DISTURBANCE (General disorders) | 1 (1) | 2 (2) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 2 (2) | 3 (4) | 2 (3)
INJECTION SITE ERYTHEMA (General disorders) | 2 (3) | 1 (1) | 1 (1)
INJECTION SITE PAIN (General disorders) | 4 (4) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 3 (4) | 3 (3) | 1 (1)
INJECTION SITE SWELLING (General disorders) | 2 (3) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 4 (4)
PAIN (General disorders) | 1 (1) | 2 (2) | 2 (3)
PERIPHERAL SWELLING (General disorders) | 3 (3) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 3 (6) | 3 (3) | 3 (4)
TEMPERATURE INTOLERANCE (General disorders) | 0 (0) | 2 (2) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 3 (4) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 4 (6) | 4 (5) | 3 (3)
CONJUNCTIVITIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
EAR INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
FUNGAL INFECTION (Infections and infestations) | 2 (4) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 3 (4) | 0 (0) | 3 (3)
GASTROENTERITIS VIRAL (Infections and infestations) | 2 (2) | 1 (1) | 1 (2)
HERPES ZOSTER (Infections and infestations) | 4 (5) | 2 (5) | 1 (1)
INFLUENZA (Infections and infestations) | 3 (3) | 4 (4) | 1 (2)
LOCALISED INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 8 (17) | 11 (20) | 7 (16)
ORAL HERPES (Infections and infestations) | 1 (1) | 3 (9) | 1 (4)
PHARYNGITIS (Infections and infestations) | 1 (3) | 2 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (2) | 1 (1) | 2 (2)
PYELONEPHRITIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 2 (3) | 8 (11) | 9 (12)
TOOTH INFECTION (Infections and infestations) | 2 (4) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 (80) | 11 (18) | 11 (24)
URINARY TRACT INFECTION (Infections and infestations) | 13 (29) | 9 (14) | 9 (19)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 1 (2)
ANIMAL BITE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 6 (9) | 1 (1) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 3 (5) | 3 (4) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 4 (5) | 3 (5) | 4 (7)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 21 (56) | 19 (60) | 16 (36)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (3)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 0 (0) | 2 (2) | 3 (3)
BLOOD PRESSURE INCREASED (Investigations) | 2 (3) | 0 (0) | 0 (0)
VITAMIN D DECREASED (Investigations) | 0 (0) | 2 (2) | 0 (0)
WEIGHT INCREASED (Investigations) | 2 (2) | 1 (2) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 (9) | 7 (7) | 9 (13)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9) | 3 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3) | 3 (3)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (7) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 5 (6)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (10) | 4 (10)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
BALANCE DISORDER (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4) | 8 (10) | 3 (3)
DYSAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 9 (17) | 12 (15) | 6 (9)
HYPOAESTHESIA (Nervous system disorders) | 4 (7) | 4 (5) | 7 (7)
LETHARGY (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
MIGRAINE (Nervous system disorders) | 3 (4) | 4 (4) | 1 (2)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 10 (11) | 5 (7) | 7 (10)
MUSCLE SPASTICITY (Nervous system disorders) | 2 (5) | 2 (2) | 5 (6)
NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 4 (8) | 3 (6) | 4 (11)
SCIATICA (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1)
SOMNOLENCE (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0)
TENSION HEADACHE (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
TREMOR (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0)
ANXIETY (Psychiatric disorders) | 6 (8) | 3 (3) | 3 (5)
DEPRESSION (Psychiatric disorders) | 4 (5) | 7 (8) | 5 (6)
INSOMNIA (Psychiatric disorders) | 4 (4) | 6 (7) | 5 (5)
PANIC ATTACK (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
HYPERTONIC BLADDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3)
MICTURITION URGENCY (Renal and urinary disorders) | 2 (2) | 3 (3) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 3 (3) | 4 (4) | 2 (2)
URINARY INCONTINENCE (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 4 (7) | 5 (6)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (3)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 6 (6)
PARANASAL SINUS DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
HAND DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
MILIARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 8 (13) | 5 (6) | 3 (3)
URTICARIA (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
HYSTERECTOMY (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3)
TOOTH EXTRACTION (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 (0) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02545868/Prot_002.pdf
  • Statistical Analysis Plan (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT02545868/SAP_000.pdf